CLINICAL TRIAL: NCT04751695
Title: Comparison of Oxidative Stress Parameters, Trace, Element and Quality of Life Levels in Healthy Men Before and After Covid-19 Vaccines
Brief Title: Oxidative Stress Parameters, Trace Element and Quality of Life in Men Before and After Covid-19 Vaccines
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Izmir Bakircay University (Other)
Collaborators: Cigli Regional Training Hospital (Other); Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Kadirhan Ozdemir, PT, PhD., Assist. Prof., Izmir Bakircay University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2021-01-174
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Covid-19 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CoronoVac Vaccine Group (Experimental)
  Interventions: Biological: CoronoVac Vaccine

INTERVENTIONS:
Biological: CoronoVac Vaccine — CoronaVac vaccines will be inoculated in 2 doses with an interval of 24 days.

SUMMARY:
With the rapid spread of COVID-19 (SARS-CoV-2) disease all over the world and the announcement of a pandemic, research on many different drug approaches has begun and these researches continue today. Although measures such as social distance, quarantine and isolation are effective in reducing the spread of SARS-CoV-2 in the short term during the pandemic, there is no effective treatment method yet. It is known that especially healthcare workers, the elderly and individuals with underlying health problems are at high risk. However, gender differences in COVID-19 clinical outcomes are thought to exist, and there is growing evidence that the disease is more severe in men than in women and mortality rates are higher.With the global consensus that the most effective approach to control the COVID-19 pandemic is a vaccination that is effective in COVID-19, vaccines have been developed with many different methods. CoronaVac vaccine (inactivated + aluminum adjuvant vaccine) is a vaccine developed with the inactive method, which is the classic vaccine production method. After the completion of Phase 1 and Phase 2 trials of the vaccine, Phase 3 trials were initiated to investigate the effectiveness of the vaccine in 4 different countries, including Turkey. Emergency use approval has been given for the CoronaVac vaccine by Turkish Pharmaceuticals and Medical Devices Agency. Researching the effects of vaccination on oxidative stress parameters, trace element and quality of life levels in COVID-19 may provide useful information in determining the effects of COVID-19 vaccine. It is thought that the anti-inflammatory and antioxidant properties of some vitamins and trace elements may be associated with positive results in COVID-19 patients, and the physiological roles of these vitamins and trace elements in COVID-19 have been demonstrated by studies. It is important to investigate the levels of free radicals known to be effective in the development of cardiovascular disease due to oxidative stress, which can provide information on determining the risk of cardiovascular complications in the COVID-19 pandemic. In addition, the quality of life of individuals decreases in the COVID-19 pandemic.This study is planned to be carried out by including male individuals to be vaccinated in İzmir Bakırçay University Çiğli Training and Research Hospital. Determination of oxidative stress parameters, trace element levels and quality of life levels before and after vaccination applications to be applied to individuals within the scope of the study; It was planned to compare these data before and after vaccination. After analyzing the data obtained from the research with appropriate statistical methods, the data will be evaluated.

DETAILED DESCRIPTION:
Coronavirus-2019 (COVID-19) is a global epidemic that has serious consequences and affects the world with its rapid spread and high mortality rate. The number of people infected with Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV2) is rapidly increasing. COVID-19 patients may have pneumonia, severe symptoms of Acute Respiratory Distress Syndrome (ARDS) and multiple organ failure, as well as cases with no symptoms.

Although social distance, quarantine and isolation are effective in reducing the spread of SARS-CoV-2 in the short term during the pandemic, there is no effective treatment method yet. It is known that especially healthcare workers, the elderly and individuals with underlying health problems are at high risk. However, gender differences in COVID-19 clinical outcomes are thought to exist, and there is growing evidence that the disease is more severe in men than in women and mortality rates are higher.

The highly contagious nature of SARS-CoV-2 has led to millions of cases worldwide, strengthening the global need for an effective vaccine to halt the spread of the disease and reduce the number of deaths. With the global consensus that the most effective approach to control the COVID-19 pandemic is a vaccination that is effective in COVID-19, many different vaccines have been tested with the acceleration of vaccination studies. According to the data of the World Health Organization, there are 236 vaccines in total, with clinical (63) and pre-clinical (173) studies developed using 10 different methods. Types of vaccines for COVID-19 include conventionally live attenuated viruses, inactivated virus protein or polysaccharide conjugated subunit vaccines, virus-like particles (VLPs), nucleic acid (DNA and RNA), viral vectors (replicating and non-replicating), and and other vaccines consisting of recombinant proteins.

Although the production of virus-based vaccines takes longer than other vaccines, the immune response is expected to be at a good level. Measles, mumps, Hepatitis A and chickenpox vaccines are examples of vaccines developed with the virus-based method. CoronaVac vaccine (inactivated + aluminum adjuvant vaccine) is a vaccine developed by the inactive method (produced and inactivated by the SARS-CoV-2 virus in the laboratory), which is the classic vaccine production method. China-based vaccine development Sinovac Biotech Ltd. Made by the biopharmaceutical company named. After the completion of Phase 1 and Phase 2 studies of the vaccine, Phase 3 studies were initiated to investigate the effectiveness of the vaccine in 4 different countries, including our country. Emergency use approval has been given for the CoronaVac vaccine by Turkish Pharmaceuticals and Medical Devices Agency.

The clinical picture of COVID-19 can be heterogeneous, ranging from asymptomatic to severe disease, which can be associated with a cytokine storm. The pathogenesis of COVID-19 is not fully understood, but is likely multifactorial and, in severe cases, with a systemic hyperinflammatory response and associated thromboembolic complications.

Some vitamins and nutrients may be beneficial for patients infected with COVID-19 due to their anti-inflammatory and antioxidant properties. Vitamins such as A, B, C, D, E and folate, and trace elements such as iron, zinc, magnesium, selenium and copper play important roles in supporting both innate and adaptive immune systems.

Free radicals are continuously formed at the active site of enzymes as intermediates in enzymatic reactions occurring during cell metabolism. Reactive oxygen species and reactive nitrogen, known as intermediates, sometimes leak from the active site of enzymes and accidentally interact with molecular oxygen and form free oxygen radicals. Lipids, proteins, enzymes, carbohydrates, and DNA can be damaged due to oxidative stress, random breaks and bonds in DNA chains may occur as a result of damage to membranes, damage to enzymes and structural proteins may result in cell death, and these phenomena may result in cancer, neurodegenerative and cardiovascular diseases, diabetes and It constitutes the molecular basis in the development of autoimmune disorders.

With the quarantine measures applied, not going out and staying at home causes the person to stay away from his daily routine life, the increase in the time spent at home, the pandemic news that is constantly being listened to and watched cause increasing anxiety, causing both changes in mood and a more sedentary life . Studies have also reported that negative psychological effects such as post-traumatic stress symptoms, confusion and anger as a result of quarantine have been reported. In addition, it has been said that restriction often causes boredom, disappointment and a feeling of isolation. These consequences, brought about by the COVID-19 pandemic, negatively affect the quality of life of individuals. During the COVID-19 pandemic, it has been reported that the depression and anxiety levels of healthcare workers increased and their quality of life decreased.

The objective of this study is to compare and determined and the changes of oxidative stress parameters, trace element and quality of life levels in healthy men just before the first dose of COVID-19 vaccine and on the 7th day after the second dose of COVID19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Agree to voluntarily participate in the study

Exclusion Criteria:

* Have been taking trace element supplements for the past 2 weeks
* Body mass index over 40 kg/m2
* Diagnosed with Covid-19 in advance
* Not diagnosed with any chronic disease

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Change of the levels of Oxidative Stress Parameter 1 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Oxidative Stress Parameter including Superoxide Dismutase (SOD) will be studied by photometric method in Medical Biochemistry Laboratory.
Change of the levels of Oxidative Stress Parameter 2 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Oxidative Stress Parameters including Malondialdehyde (MDA) will be studied by photometric method in Medical Biochemistry Laboratory.
Change of the levels of Oxidative Stress Parameter 3 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Oxidative Stress Parameter including Total Antioxidant Level (TAL) will be studied by photometric method in Medical Biochemistry Laboratory.
Change of the levels of Oxidative Stress Parameter 4 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Oxidative Stress Parameters including Total Oxidant Level (TOL) will be studied by photometric method in Medical Biochemistry Laboratory.
Change of the levels serum trace element 1 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace element including zinc levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method
Change of the levels serum trace element 2 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace elements including selenium levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels serum trace element 3 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace element including potassium levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels serum trace element 4 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace element including sodium levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels serum trace element 5 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace elements including calcium levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels serum trace element 6 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace element including magnesium levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels serum trace element 7 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace element including copper levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels of quality of life | Immediately before the first dose and 4 weeks later
  SF-36 Quality of Life Scale will be used to determine the quality of life level. The scale that patients can apply themselves and in a short time; It consists of 36 items and 8 subsections. These sections are physical functionality, social functionality, role restrictions due to physical problems, role restrictions due to emotional problems, pain, energy level / vitality / vitality, mental health, and general health perception (40). The last 4 weeks are considered in the evaluation of the scale. The scale gives a separate total score for each subsection. The points obtained from the subsections are not added up. Subdivisions rate health from 0 to 100. While it expresses bad health status as "0 points", it refers to good health status as "100 points".

CONTACTS AND LOCATIONS:
Locations (1):
- Kadirhan Ozdemir, Izmir, Turkey (Türkiye)